CLINICAL TRIAL: NCT00237731
Title: Pre-hospital Morphine Titration : Comparison of 0,05 Versus 0,1 mg/kg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Roques, UHToulouse
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0505103
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Severe, Acute Pain in a Pre-hospital Setting
Keywords: Acute pain; Morphine titration; Analgesia; Pre-hospital care
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): morphine 0.05
  Interventions: Drug: morphine
- 2 (Active Comparator): morphine 0.10
  Interventions: Drug: morphine

INTERVENTIONS:
Drug: morphine — morphine 0.05
  Arms: 1
Drug: morphine — morphine 0.10
  Arms: 2

SUMMARY:
Efficacy and safety of morphine titration on acute pain in emergency medical mobile units with initial bolus of 0.1 mg/kg plus 0.05 mg/kg versus morphine titration with initial bolus of 0.05 mg/kg plus 0.025 mg/kg

DETAILED DESCRIPTION:
STUDY OBJECTIVE : Assess the efficacy of a morphine dose of 0.1 mg/kg versus a morphine dose of 0.05 mg/kg in pre-hospital pain METHODS : Consecutive patients with severe, acute pain defined as a verbal rating scale (VRS) of 60/100 or higher may be included. 106 patients at all are required in the study. They will be randomised in two groups : group A will receive an initial intravenous injection of 0.05 mg/kg then injections of 0.025 mg/kg every 5 minutes and group B will receive an initial intravenous injection 0.1 mg/kg then injections of 0.05 mg/kg every 5 minutes. The pain scale will be checked every 5 minutes during 30 minutes. The titration will be stopped before, if the VRS is < or = 30. The patient will be followed during the study until 60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Severe, acute pain defined by a VRS of 60/100 or higher
* Male or female over 18 years
* Cared by a medical emergency care unit
* Written informed consent
* Affiliated to social security

Exclusion Criteria:

* A known opioid or paracetamol hypersensitivity
* Patient not agree ta participate at the study
* Pregnancy
* Uncontrolled epilepsia
* Incapacity to understand the VRS
* Renal, respiratory, or liver disease
* Patients who have received sedative drugs or alcohol (< 6h)
* Acute respiratory, haemodynamic or neurologic failure
* Patients who have already received an analgesic (< 6h)
* Drug addiction
* Patients under protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2005-09; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
A verbal rating scale of 30/100 or lower measured 30 minutes after initial administration

SECONDARY OUTCOMES:
Time to obtain an analgesia, defined by a VRS < or = 30
Patients' satisfaction with analgesia (pain relief classified as excellent, good, mild or weak)
Investigators' satisfaction with analgesia (pain relief classified as excellent, good, mild or weak)
Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis DUCASSE, Principal Investigator — University Hospital, Toulouse, France
Locations (1):
- SAMU 31 Hôpital PURPAN, Toulouse, France

REFERENCES:
- [Background] Ricard-Hibon A, Leroy N, Magne M, Leberre A, Chollet C, Marty J. [Evaluation of acute pain in prehospital medicine]. Ann Fr Anesth Reanim. 1997;16(8):945-9. doi: 10.1016/s0750-7658(97)82142-9. French. PMID 9750642
- [Background] Ricard-Hibon A, Marty J. Prise en charge de la douleur en milieu préhospitalier, In SFAR, Conférences d'actualisation 2001, Paris, Elsevier,2001;pp 709-22
- [Background] SFAR. Quelles sont les modalités de réalisation d'une sédation et/ou d'une analgésie du malade en ventilation spontanée. In : SFAR eds. Modalités de la sédation et/ou de l'analgésie en situation extrahospitalière : Conférence d'experts. Paris, Elsevier;2000;pp 37-51
- [Background] SFUM. Troisième conférence de consensus en médecine d'urgence de la Société francophone d'urgence médicale. Le traitement médicamenteux de la douleur de l'adulte dans un service d'accueil et d'urgence. Réan Urg 1993; 2:321-7
- [Result] Bounes V, Charpentier S, Houze-Cerfon CH, Bellard C, Ducasse JL. Is there an ideal morphine dose for prehospital treatment of severe acute pain? A randomized, double-blind comparison of 2 doses. Am J Emerg Med. 2008 Feb;26(2):148-54. doi: 10.1016/j.ajem.2007.04.020. PMID 18272093
- See also: Observatoire Régional Urgences Midi-Pyrénées, Rapport annuel sur l'activité des services d'urgence 2004 — http://www.orumip.fr